CLINICAL TRIAL: NCT03878979
Title: Preoperative Immune Checkpoint Inhibitor Therapy for Patients With Primary Untreated or Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck (RM-SCCHN)
Brief Title: Preoperative Immune Checkpoint Inhibitor for Patients With Primary Untreated or Recurrent/Metastatic SCCHN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: J1923; IRB00207577 (Other: JHM IRB); CA209-9H7 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Head and Neck Cancer; Head and Neck Cancer Metastatic
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Nivolumab; MD1

STUDY DESIGN:
Intervention Model Description: The study will accrue to 2 cohorts, each of which consists of about 12 patients. If enrollment on 1 cohort is significantly faster, the lesser enrolling cohort number of patients may be decreased in favor of the better enrolling cohort to keep the total number of evaluable patients at 24 patients.Total of 24 patients will be accrued to the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Newly diagnosed SCCHN (Experimental): One dose of nivolumab given about 4 weeks before surgical resection (removal) of a newly diagnosed SCCHN.
  Interventions: Drug: Nivolumab 480mg and surgical resection
- Recurrence of SCCHN (Experimental): One dose of nivolumab given about 4 weeks before surgical resection (removal) of SCCHN which has recurred.
  Interventions: Drug: Nivolumab 480mg and surgical resection

INTERVENTIONS:
Drug: Nivolumab 480mg and surgical resection — One dose of Nivolumab 480mg given four weeks prior to surgical resection.
  Other Names: Opdivo; Ono Pharmaceutical (ONO) 4538; BMS-936558; Medarex Incorporated (MDX) 1106

SUMMARY:
Nivolumab, also known as (Bristol Myers Squibb (BMS)) BMS-936558, before surgery to people with newly diagnosed or recurrent squamous cell carcinoma of head and neck (SCCHN).

DETAILED DESCRIPTION:
This research is being done to see if it is safe and feasible to give the investigational drugs, nivolumab (also known as BMS-936558) before surgery to people with newly diagnosed or recurrent squamous cell carcinoma of head and neck (SCCHN). Patients with recurrent disease may have a limited number of sites of metastatic (spread) squamous cell carcinoma of head and neck. Another goal of this study is to learn how nivolumab impacts the immune system's ability to treat the cancer. While nivolumab is approved by the U. S. Food and Drug Administration (FDA) for the treatment of patients with metastatic SCCHN with progression on or after platinum-based chemotherapy, the word "investigational" in this context means that the study drugs are not approved by the FDA for the treatment of head and neck cancers prior to surgery and thus is still being tested in research studies. However, the FDA is allowing the use of nivolumab in this study.

This study will have two arms. Cohort (arm) 1 will examine one dose of nivolumab given about 4 weeks before surgical resection (removal) of a newly diagnosed SCCHN. Twelve patients will be enrolled to this arm. Cohort 2 will examine one dose of nivolumab given about 4 weeks before surgical resection (removal) of SCCHN which has recurred and possibly spread to distant sites, but still can be resected with one surgery. Twelve patients will be enrolled to this arm.

ELIGIBILITY:
Inclusion:

Cohort 1: Subjects must have histologically confirmed previously untreated squamous cell carcinoma of the head and neck which is amenable to surgical resection as part of standard of care.

Cohort 2: Subjects must have histologically confirmed recurrent squamous cell carcinoma of head and neck, which is amenable for salvage surgery. Sites of recurrence may either be locoregional or distant if resection can be done ideally in one surgical field.

* The primary site should be a head and neck squamous cell carcinoma (including, but not limited to oral cavity, oropharynx, hypopharynx, or larynx, paranasal sinuses, nasal cavity). Squamous cell carcinoma of unknown primary, diagnosed in lymph nodes in neck, can be included but should be tested for p16 and confirmed specific assay.
* Subjects with oropharyngeal primary tumors must have confirmation of human papillomavirus (HPV) tumor status per clinical standards, although not necessary at enrollment.
* Subjects must have been determined to be candidates for surgical resection by a multidisciplinary team including a surgeon, a medical oncologist and a radiation oncologist.
* Subjects must have at least one lesion that can be biopsied at baseline.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
* Age >18 years.
* Life expectancy of greater than 6 months.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes ≥ 1,500/ microliter (mcL)
  * absolute neutrophil count ≥ 1,000/mcL
  * platelets ≥ 100,000/mcL
  * total bilirubin ≤ 1.5 X institutional upper limit of normal (except subjects with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL)
  * aspartate aminotransferase (AST) (SGOT) / alanine aminotransferase (ALT) (SGPT) ≤ 3 X institutional upper limit of normal
  * Creatinine OR creatinine clearance within normal institutional limits OR ≥ 40 mL/min (using modified Cockcroft-Gault formula) for patients with creatinine levels above institutional normal.
* Resting and walking O2 saturation must remain above 90% at the time of screening
* Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment.
* Women must not be breastfeeding
* Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatment and for 5 months post-treatment completion. Women should use an adequate method(s) of contraception (Refer to nivolumab Investigator's Brochure (IB) for WOCBP and methods of contraception to be provided)
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception (Refer to protocol appendix E) for the duration of treatment with study treatment(s) and 7 months post-treatment completion. In addition, male participants must be willing to refrain from sperm donation during this time. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception
* Patient understands the study regimen, its requirements, risks and discomforts and is able and willing to sign the informed consent form. Voluntary signed and dated Institutional Review Board (IRB) / Independent Ethics Committee (IEC) approved written informed consent form in accordance with regulatory and institutional guidelines must be obtained before the performance of any protocol related procedures that are not part of normal patient care. Subjects must be competent to report adverse events (AEs), understand the drug dosing schedule and use of medications to control AEs.
* Measurable disease - either radiologically (per RECIST) or clinically measurable on exam in order to assess treatment response.

Exclusion Criteria

* Any active history of a known autoimmune disease. Subjects with vitiligo, type 1 diabetes mellitus, residual hypothyroidism requiring hormone replacement, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Patients who have had prior chemotherapy for newly diagnosed (cohort 1) or recurrent (cohort 2) head and neck cancer. In cohort 2 only, previous perioperative chemotherapy or chemoradiation for the management of localized or locally advanced disease permitted.
* Patients who had prior surgical resection of distant metastasis (metastasectomy) within 3 months of enrollment.
* Patients who received prior therapy with anti-programmed death (PD) 1 (anti-PD-1), anti-PD-L1, anti-PD-L2, cluster of differentiation (CD)137 (CD137), anti-cytotoxic T-lymphocyte associated (CTLA) protein 4 (anti-CTLA-4) (cytotoxic T-lymphocyte associated protein 4) antibody therapies, any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways. Any live / attenuated vaccine (eg varicella, zoster, yellow fever, rotavirus, oral polio and measles, mumps, rubella (MMR)) during treatment and until 100 days post last dose.
* Patients with uncontrolled brain metastases
* Patients with brain metastases must have stable neurologic status following local therapy (surgery or radiation) for at least 2 weeks without the use of steroids or on stable or decreasing dose of < 10mg daily prednisone (or equivalent), and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with a history of carcinomatous meningitis are not eligible.
* Patients who have an active concurrent malignancy that is not controlled/cured and could impact life expectancy within the next 3 years. E.g. patients with localized cutaneous squamous cell carcinoma or basal cell carcinoma or treated prostate cancer with no evidence of disease progression may be allowed to enroll after review by the study team.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, administration of live vaccination in the prior 3 months, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, myocardial infarction or new onset angina within six months of enrollment, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women who are pregnant or nursing.
* Men with female partners who are not willing to use contraception.
* Active infection with hepatitis B or hepatitis C.
* Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids and adrenal replacement steroid doses < 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Patients Epstein-Barr virus + (EBV+) with nasopharynx carcinoma
* Patient with HIV are excluded given the unknown risk of interaction with HAART and the unknown benefit of immunotherapy in this population.
* Participants who have received a live / attenuated vaccine within 30 days of first treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanguy Lim-Seiwert, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Reccurence of SCCHN: One dose of nivolumab given about 4 weeks before surgical resection (removal) of SCCHN which has recurred.
  Nivolumab 480mg and surgical resection: One dose of Nivolumab 480mg given four weeks prior to surgical resection.
Period: Overall Study
Arm/Group | Newly Diagnosed SCCHN | Reccurence of SCCHN
Started | 20 | 6
Completed | 20 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Newly Diagnosed SCCHN | Reccurence of SCCHN | Total
Number analyzed (Participants) | 20 | 6 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 11
  >=65 years | 13 | 2 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 8
  Male | 13 | 5 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 16 | 4 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 6 | 26

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by Number of Participants With Drug-related Adverse Events
Description: Safety of neoadjuvant nivolumab administration in patients with newly diagnosed head and neck cancer and those with locoregional recurrence or oligometastatic disease undergoing surgical resection measured by number of participants with drug related adverse events as defined by CTCAE v5.0, occurring up to 100 days after the last dose of nivolumab or 30 days after surgery (whichever is longer)
Time Frame: Up to 100 days after the last dose of nivolumab or 30 days after surgery, whichever is longer (up to 100 days per participant)
Measure: Count of Participants; unit: Participants
Arm/Group | Newly Diagnosed SCCHN | Reccurence of SCCHN
Number analyzed (Participants) | 20 | 6
Participants | 19 | 2

2. Primary Outcome: Feasibility as Measured by Number of Participants With Successful Completion of Preoperative Treatment and no Extended Treatment-related Delays
Description: Feasibility of neoadjuvant nivolumab administration in patients with newly diagnosed head and neck cancer and those with locoregional recurrence or oligometastatic disease undergoing surgical resection, measured by number of participants with successful completion of preoperative treatment and proceeding to surgery without any extended treatment related delays more than > 28 days from pre-planned day 0.
Time Frame: Up to 100 days after the last dose of nivolumab or 30 days after surgery (whichever is longer per participant)
Measure: Count of Participants; unit: Participants
Arm/Group | Newly Diagnosed SCCHN | Recurrence of SCCHN
Number analyzed (Participants) | 20 | 6
Participants | 20 | 6

3. Secondary Outcome: Major Pathologic Response Rate
Description: Number of participants with < 10% residual tumor in the resection specimen.
Time Frame: Day 0 (Surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Newly Diagnosed SCCHN | Reccurence of SCCHN
Number analyzed (Participants) | 19 | 4
Participants | 3 | 2

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Number of months until radiologic or clinical progression or death, whichever occurs first.
Time Frame: up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Newly Diagnosed SCCHN | Reccurence of SCCHN
Number analyzed (Participants) | 20 | 6
months | NA [NA to NA] — not estimable due to small number of PFS events | 23 [11.5 to NA] — not estimable due to small number of PFS events

5. Secondary Outcome: Radiographic Response Rate
Description: Number of participants with response as determined by RECIST version 1.1 and immune-related response criteria (irRC). Per RECIST criteria, Complete response (CR) is a disappearance of all target lesions, Partial response (PR) is >= 30% decrease in the sum of the largest diameter (LD) of target lesions, Progressive disease (PD) is >= 20% increase in the sum of the LD of target lesions.
  Per irRC, immune-related Complete Response (irCR) is the disappearance of all lesions, measured or unmeasured, and no new lesions; an immune-related Partial Response (irPR) is a 50% drop in tumour burden from baseline as defined by the irRC; and immune-related Progressive Disease (irPD) is a 25% increase in tumour burden from the lowest level recorded.
Time Frame: up to 4 weeks after the last dose of nivolumab
Population: Overall number of participants analyzed for newly diagnosed (15) is different than the number who started in participant flow (20), because 5 patients did not have measurable disease at baseline.
  Overall number of participants analyzed for recurrence (5) is different than the number who started in participant flow (6), because 1 patient visit was not done.
Measure: Count of Participants; unit: Participants
Arm/Group | Newly Diagnosed SCCHN | Recurrence of SCCHN
Number analyzed (Participants) | 15 | 5
Participants
  Partial Response (PR) | 1 | 1
  Complete Response (CR) | 0 | 0
  Stable Disease (SD) | 9 | 2
  Progressive Disease (PD) | 4 | 2
  Not evaluable | 1 | 0

ADVERSE EVENTS:
Time Frame: approximately 3 years 3 months
Arm/Group | Newly Diagnosed SCCHN | Reccurence of SCCHN
All-Cause Mortality (participants affected / at risk) | 4/20 | 1/6
Serious Adverse Events (participants affected / at risk) | 5/20 | 0/6
Other Adverse Events (participants affected / at risk) | 20/20 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Newly Diagnosed SCCHN (N=20) | Reccurence of SCCHN (N=6)
Cardiac ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Fever (Immune system disorders) | 1 (1) | 0 (0)
Left arm edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Newly Diagnosed SCCHN (N=20) | Reccurence of SCCHN (N=6)
Abdominal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abrasion on chin (General disorders) | 1 (1) | 0 (0)
Achy bilateral leg muscles (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anemia (Cardiac disorders) | 4 (4) | 0 (0)
Anorexia (Psychiatric disorders) | 2 (2) | 0 (0)
Bilateral hand tremor (Nervous system disorders) | 1 (1) | 0 (0)
Bilateral shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Blood and lymphatic system disorders-other (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bruising left hand (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Chronic arthritis (Immune system disorders) | 0 (0) | 1 (1)
Concentration impairment with increase in gabapentin (Psychiatric disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Coughing in morning (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decreased absolute lymphocyte count (Investigations) | 2 (2) | 2 (2)
Decreased lymphocyte count (Investigations) | 1 (1) | 0 (0)
Decreased mean platelet volume (Investigations) | 0 (0) | 1 (1)
Decreased range of motion - neck (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Distal tip of incision has necrosis (Surgical and medical procedures) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Dysphagia (Nervous system disorders) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Elevated alanine aminotransferase (Investigations) | 1 (1) | 0 (0)
Elevated alk (Investigations) | 1 (1) | 0 (0)
Elevated alkaline phosphatase (Investigations) | 1 (1) | 0 (0)
Elevated alt (Investigations) | 1 (1) | 0 (0)
Elevated aspartate aminotransferase (Investigations) | 1 (1) | 0 (0)
Elevated tsh (Endocrine disorders) | 1 (1) | 0 (0)
Eyelid-drooping (Eye disorders) | 1 (1) | 0 (0)
Facial edema (right side) (General disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 2 (2) | 0 (0)
Facial pain (left jaw) worsening (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Facial pain (right side jaw) (General disorders) | 1 (1) | 0 (0)
Fatigue (Nervous system disorders) | 4 (4) | 1 (1)
Fever of 101.5 f (General disorders) | 0 (0) | 1 (1)
Floaters right eye (Eye disorders) | 1 (1) | 0 (0)
Forgetfulness (Nervous system disorders) | 1 (1) | 0 (0)
Gait imbalance (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Generalized muscle aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Halitosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 2 (2) | 1 (1)
Headache (consistent) (General disorders) | 1 (1) | 0 (0)
Headache behind both eyes (General disorders) | 1 (1) | 0 (0)
Headache in back of eye going to back of head (General disorders) | 1 (1) | 0 (0)
Hematoma in left eye (Eye disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Increased fatigue (General disorders) | 1 (1) | 0 (0)
Increased pain and swelling of gums and mouth (General disorders) | 1 (1) | 0 (0)
Increased pain with swallowing (Gastrointestinal disorders) | 1 (1) | 0 (0)
Influenza b infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0)
Intermittent dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Intermittent facial pain (right side jaw) (General disorders) | 1 (1) | 0 (0)
Intermittent sternal pain (deep inspiration) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intermittent urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Jaw pain (facial pain) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Left arm bruise (General disorders) | 1 (1) | 0 (0)
Left ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Left face & neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Left lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Left peri-oral numbness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Left shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leukocytosis (Immune system disorders) | 0 (0) | 1 (1)
Light headedness (Nervous system disorders) | 1 (1) | 0 (0)
Light sensitivity (Eye disorders) | 1 (1) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (2)
Lymphocytes absolute decreased (Investigations) | 1 (1) | 0 (0)
Maculopapular rash - (chest) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Maculopapular rash-lower back (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0)
Memory impairment with increase in gabapentin (Nervous system disorders) | 1 (1) | 0 (0)
Mild depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mild nausea (General disorders) | 1 (1) | 0 (0)
Mild shortness of breath (stair climbing) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mild swelling in the area of tumor (General disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Necrosis & dehiscence (Surgical and medical procedures) | 0 (0) | 1 (1)
Numbness - thumb and first 2 fingers (Nervous system disorders) | 1 (1) | 0 (0)
Numbness (right side face) (Nervous system disorders) | 1 (1) | 0 (0)
Numbness in left neck area (Nervous system disorders) | 1 (1) | 0 (0)
Numbness/left side of face (Nervous system disorders) | 1 (1) | 0 (0)
Occasional cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Occasional diarrhea following laxative use (Gastrointestinal disorders) | 1 (1) | 0 (0)
Occasional lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Occasional mild nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Occasional nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
Pain bi-lateral forearm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Paresthesia on left side face (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (left ear) (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (numbness in fingertips bilaterally) (Nervous system disorders) | 0 (0) | 1 (1)
Pedal edema (General disorders) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia (lung infection) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Post-surgical mouth pain (Surgical and medical procedures) | 1 (1) | 0 (0)
Post-surgical neck pain (Surgical and medical procedures) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Right shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Right sided ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Right sided headache (General disorders) | 1 (1) | 0 (0)
Significant pain in right ear (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Skin infection (left great toe cellulitis) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Small reddened area- right upper arm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Soreness in left neck (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Syncope (during blood draw) (Nervous system disorders) | 1 (1) | 0 (0)
Taste alteration (dysgeusia) (Nervous system disorders) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Visual changes in left eye (Eye disorders) | 1 (1) | 0 (0)
Voice changes (hoarseness) (General disorders) | 1 (1) | 0 (0)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Weight loss (General disorders) | 2 (2) | 0 (0)
Worsening constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Worsening fatigue (Nervous system disorders) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Oral pain (tongue) (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT03878979/Prot_SAP_000.pdf